CLINICAL TRIAL: NCT00869960
Title: Impact of Menstrual Cycle on Antiretroviral Pharmacokinetics in Healthy Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: F080428014; 1K23AI074390-01A2 (NIH)
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Results first posted 2012-04-12 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — Tenofovir; Emtricitabine; Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antiretroviral therapy (Experimental): Healthy volunteers received two doses of Tenofovir, Emtricitabine, Atazanavir and Ritonavir administered twice (on day 6 - 10 and day 20 - 25 after day of Follicular phase); with pharmacokinetic measurements at 6 - 10 days after menses and then again at day 20 - 25 after menses.
  Interventions: Drug: tenofovir; Drug: emtricitabine; Drug: atazanavir; Drug: ritonavir

INTERVENTIONS:
Drug: tenofovir — tenofovir 300 mg one dose on 2 separate visits: within 5 days after Day 1 of Follicular phase and then within a 4 day window of the leutal phase (day 14 of the menstrual cycle)
Drug: emtricitabine — emtricitabine 200 mg on 2 separate visits: within 5 days after Day 1 of Follicular phase and then within a 4 day window of the leutal phase (day 14 of the menstrual cycle).
Drug: atazanavir — atazanavir 300mg one dose on 2 separate visits: within 5 days after Day 1 of Follicular phase and then within a 4 day window of the leutal phase (day 14 of the menstrual cycle).
Drug: ritonavir — ritonavir 100 mg one dose on 2 separate visits: within 5 days after Day 1 of Follicular phase and then within a 4 day window of the leutal phase (day 14 of the menstrual cycle).

SUMMARY:
Data suggest that women taking drugs to treat human immunodeficiency virus (HIV) have higher amounts of drugs in their body compared with men taking the same dose of anti-HIV drugs. The reason for this higher drug exposure has not been determined. The primary purpose of this study is to examine whether the pharmacokinetics (factors that determine the amount of drug in the body) of anti-HIV drugs change during different phases of the menstrual cycle in women and ultimately result in higher amounts of drug in the body compared with men. In other words, we plan to examine whether changes in sex hormones throughout the menstrual cycle affect the amount of anti-HIV drugs in women. The antiretroviral drugs atazanavir, ritonavir, tenofovir and emtricitabine will be studied. This study will be conducted in healthy women since HIV may change the pharmacokinetics of anti-HIV drugs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, HIV negative, nonsmoking females between 21 and 40 years of age.
* Subjects must be within 20% of their ideal body weight and have a regular menstrual cycle, defined as at least 10 cycles per year occurring approximately every 28 ± 4 days and cycle length varying by not more than 7 days.
* Subjects must be willing and able to provide written informed consent.
* Subjects cannot be breast feeding, pregnant or be taking hormonal contraception within 3 months prior to study enrollment. However, they must agree to use an effective non-hormonal method of contraception during the study.

Exclusion Criteria:

* Subjects receiving prescription or over-the-counter products which may interact with the study medication will be excluded from the study.
* Subjects with a Grade 3 or higher laboratory liver, renal or hematology abnormality as specified below in accordance with the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table) Version 1.0, Dec 2004, will be excluded.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R. King, PharmD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Antiretroviral Therapy: Healthy volunteers
Period: Overall Study
Arm/Group | Antiretroviral Therapy
Started | 24
Completed | 22
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Combination Antiretroviral Therapy: Single dose administration of tenofovir, emtricitabine, atazanavir and ritonavir to healthy women
Arm/Group | Combination Antiretroviral Therapy
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Tenofovir Systemic Exposure During the Follicular Phase (Days 6-10 After Menses)
Description: Systemic exposure determined by area under the concentration time curve was measured by blood drawn for PK assessment at the following times: 0 (time of dose), 0.5, 1, 2, 4,6, 8, 12 and 24 hours. The Follicular phase starts on day 1 of the menstrual cycle when estrogen and progesterone levels are lowest. this lasts 14 days. Dose administration and PK would have been drawn on day 6, 7, 8, 9, or 10 after Day 1 (start of Follicular phase).
Time Frame: between time of dosing to 24 hours after dose administered
Population: The number was determined based upon the those women who completed the study.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Antiretroviral Therapy
Number analyzed (Participants) | 22
mg*h/L | 2.4 (1.1)

2. Primary Outcome: Tenofovir Systemic Exposure During the Luteal Phase (Days 20-25 After Menses)
Description: Systemic exposure determined by area under the concentration time curve was measured by blood drawn for PK assessment at the following times: 0 (time of dose), 0.5, 1, 2, 4,6, 8, 12 and 24 hours. The Luteal phase starts on day 14 of the menstrual cycle when estrogen and progesterone levels are beginning to increase. This lasts 14 days or until Day 1 of the Follicular phase. Dose administration and PK during the Luteal phase, would have been drawn on day 20, 21, 22, 23, 24 and 25 start of Follicular phase).
Time Frame: between time of dosing tp 24 hours after dose administration
Population: The number was determined based upon the those women who completed the study.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Antiretroviral Therapy
Number analyzed (Participants) | 22
mg*h/L | 2.2 (0.07)

3. Primary Outcome: Emtricitabine Systemic Exposure During the Follicular Phase (Days 6-10 After Menses)
Description: as for outcome 1
Time Frame: Between time of dosing to 24 hours after dose administration
Population: The number was determined based upon the those women who completed the study.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Antiretroviral Therapy
Number analyzed (Participants) | 22
mg*h/L | 11.2 (4.4)

4. Primary Outcome: Emtricitabine Systemic Exposure During the Luteal Phase (Days 20-25 After Menses)
Description: as for outcome 2
Time Frame: Between time of dosing to 24 hours after dose administration
Population: The number was determined based upon the those women who completed the study.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Antiretroviral Therapy
Number analyzed (Participants) | 22
mg*h/L | 10.2 (3.7)

5. Primary Outcome: Atazanavir Systemic Exposure During the Follicular Phase (Days 6-10 After Menses)
Description: as for outcome 1
Time Frame: Between time of dosing to 24 hours after dose administration
Population: The number was determined based upon the those women who completed the study.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Antiretroviral Therapy
Number analyzed (Participants) | 22
mg*h/L | 23.9 (13.5)

6. Primary Outcome: Atazanavir Systemic Exposure During the Luteal Phase (Days 20-25 After Menses)
Description: as for outcome 2
Time Frame: Between time of dosing to 24 hours after dose administration
Population: The number was determined based upon the those women who completed the study.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Antiretroviral Therapy
Number analyzed (Participants) | 22
mg*h/L | 22.4 (9.1)

7. Primary Outcome: Ritonavir Systemic Exposure During the Follicular Phase (Days 6-10 After Menses)
Description: as for outcome 1
Time Frame: Between time of dosing to 24 hours after dose administration
Population: The number was determined based upon the those women who completed the study.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Antiretroviral Therapy
Number analyzed (Participants) | 22
mg*h/L | 7.2 (3.6)

8. Primary Outcome: Ritonavir Systemic Exposure During the Luteal Phase (Days 20-25 After Menses)
Description: as for outcome 2
Time Frame: Between time of dosing to 24 hours after dose administration
Population: The number was determined based upon the those women who completed the study.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Antiretroviral Therapy
Number analyzed (Participants) | 22
mg*h/L | 6.7 (3.1)

ADVERSE EVENTS:
Arm/Group | Antiretroviral Therapy
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No